CLINICAL TRIAL: NCT06161727
Title: Detection and Prevalence of Human Papillomavirus (HPV) in Seminal Plasma and/or on Sperm in Men Undergoing Treatment With IVF/ICSI in Southwestern Sweden: a Prospective Study.
Brief Title: Detection and Prevalence of Human Papillomavirus (HPV) in Seminal Plasma and/or on Sperm in Men Undergoing Treatment With IVF/ICSI.
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Panagiotis Tsiartas, MD, PhD, Senior Consultant, M.D., Ph.D., Vastra Gotaland Region
Other Study IDs: SpermHPV
Record Dates: First submitted 2023-11-28; First posted 2023-12-08 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Human Papilloma Virus; Infertility, Male
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — HPV DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men with HPV-positive (HPV+) semen samples
  Interventions: Other: HPV exposure
- Men with HPV-negative (HPV-) semen samples
  Interventions: Other: HPV exposure

INTERVENTIONS:
Other: HPV exposure — According to group descriptions

SUMMARY:
This observational study aims to investigate the presence of HPV DNA in semen samples from men undergoing in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) treatment. It focuses on understanding the impact of HPV on male fertility and embryo development following IVF/ICSI. The primary goal is to determine the prevalence of HPV-positive (HPV+) semen samples among men seeking infertility treatment with IVF/ICSI. Additionally, the study aims to compare semen characteristics between HPV-positive and HPV-negative (HPV-) samples and assess the embryological outcomes after IVF/ICSI in these two groups.

Participants in this study will include men receiving IVF/ICSI treatment and providing fresh ejaculated sperm at Sahlgrenska University Hospital in Gothenburg, Sweden, over one year. Those undergoing treatments with surgically extracted sperm, sperm freezing for fertility preservation, or planning treatments involving preimplantation genetic testing or egg donation will be excluded.

The study will involve analyzing HPV DNA in semen samples through PCR, utilizing the most effective method for HPV DNA detection previously identified in a pilot study. Sperm samples collected during infertility investigations and IVF/ICSI treatments will undergo gradient centrifugation to separate different components. A portion of the sperm sample will be preserved for PCR analysis to detect HPV DNA, while the rest will be used for IVF/ICSI procedures. The results from the PCR analyses will be correlated with semen characteristics and the outcomes of IVF/ICSI treatment. Furthermore, the samples will be stored for potential future analyses related to HPV-related biomarkers for up to 5 years at Biobank.

DETAILED DESCRIPTION:
Infection with the human papillomavirus (HPV) represents one of the most widespread sexually transmitted diseases, affecting both genders. Over 100 types of HPV can cause infections in the skin or mucous membranes and are typically transmitted through skin-to-skin contact, vaginal or anal intercourse, as well as oral sex. Statistics indicate that between 50 and 80 percent of sexually active adults will experience genital HPV infections during their lifetime. These infections tend to be persistent, especially in men. Although most HPV infections are asymptomatic, they can lead to genital warts, dysplasia, cancer, infertility, and may impact the outcomes of in vitro fertilization (IVF). Despite extensive research on HPV-related conditions in women, there has been limited attention given to HPV-related conditions in men.

A systematic review and meta-analysis conducted in 2017, comprising 31 studies, revealed that the prevalence of HPV DNA in semen samples among men in the general population was 11.4%, rising to 20.4% among men with infertility. It remains unclear whether HPV localizes in seminal plasma or in cellular fractions of semen samples (such as sperm, epithelial cells, or leukocytes). Recent evidence has shown that HPV DNA can be found on the surface of sperm by binding to specific glycosaminoglycans (GAGs), such as syndecan-1, along the equatorial region of the sperm head. Additionally, a few in vitro studies have indicated that HPV DNA can be found inside sperm when mixed with the HPV virus. The potential effects of HPV on fertility are not yet fully understood. The presence of HPV infection in sperm has been associated with impaired sperm parameters, mainly sperm motility, and increased sperm DNA fragmentation. Existing evidence suggests a negative effect of HPV DNA in seminal plasma and/or on sperm on the number of live births and ongoing pregnancies, although the level of evidence remains limited. Considering that sperm is utilized in IVF, it is crucial to investigate the presence of HPV in seminal plasma and sperm in these men, as well as any potential consequences on embryo development following IVF.

The primary objective of this study is to assess the prevalence of HPV DNA in seminal plasma and/or on sperm in men undergoing in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) treatments. Furthermore, the study aims to characterize semen parameters in men with HPV-positive (HPV+) and HPV-negative (HPV-) semen samples and analyze the embryological outcomes after IVF/ICSI in men with HPV+ semen samples compared to men with HPV- semen samples.

The secondary objectives include evaluating semen parameters such as volume, sperm concentration, and motility to determine if there are differences between men with HPV+ and HPV- semen samples. Additionally, the study aims to investigate whether the embryological outcome (fertilization rate, number of high-quality embryos) after IVF/ICSI treatment differs between men with HPV+ and HPV- semen samples.

Analyses of HPV DNA in seminal plasma and/or on sperm will be conducted using the method that has demonstrated the highest performance in detecting HPV DNA, based on a previously conducted pilot study. Sperm samples are typically provided at the Fertility Laboratory at the Department of Reproductive Medicine, SU, in conjunction with infertility investigations and IVF/ICSI treatments. Usually, up to 2 mL of ejaculated sperm sample undergo gradient centrifugation, separating motile sperm from seminal plasma, immotile sperm, squamous epithelial cells, leukocytes, and bacteria. A portion of the pellet containing motile sperm is used to analyze sample parameters, primarily concentration and motility. During IVF/ICSI treatments, parts of the sperm sample are utilized for egg fertilization while the remainder is discarded. Following gradient centrifugation, sperm samples are diluted with a preservation liquid (ThinPrep®, 1:2) and stored in a refrigerator for transport to the Clinical Microbiology Department (virological laboratory) at SU (once per week) for polymerase chain reaction (PCR) analysis. ThinPrep® is routinely used to preserve and fix cell samples for HPV analysis in women. In this study, the portion of the sperm sample typically discarded and not used for IVF treatment will be utilized for HPV DNA analysis using PCR. PCR is the method routinely employed at the Clinical Microbiology Department (virological laboratory) at SU for HPV DNA detection in cervical cell samples. Results from these analyses will be correlated with sample parameters and the embryological outcome following completed IVF/ICSI treatment. Once analyzed by PCR and upon the availability of material, the samples will be stored for 5 years at Biobank Väst for potential future analyses of HPV-related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Over the course of one year, the study will include men undergoing infertility treatment with IVF/ICSI and fresh ejaculated sperm at Sahlgrenska University Hospital (SU), Gothenburg, Sweden.

Exclusion Criteria:

* Men undergoing IVF/ICSI treatments with surgically extracted sperm.
* Men undergoing sperm freezing for fertility preservation purposes or possessing previously frozen sperm.
* Sperm donors.
* Men for whom treatment with preimplantation genetic testing (PGT) or egg donation is planned.

Ages: 18 Years to 60 Years | Sex: Male
Age Groups: Adult
Study Population: Men undergoing infertility treatment with IVF/ICSI and fresh ejaculated sperm at Sahlgrenska University Hospital (SU), Gothenburg, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of HPV+ sperm samples | January 2023-March 2024
  Number of HPV + sperm samples among all recruited men undergoing infertility treatment with IVF/ICSI

SECONDARY OUTCOMES:
Semen volume in mL | January 2023-March 2024
  Is semen volume different between men with HPV+ and HPV- semen samples?
Sperm concentration in number of spermatozoa/mL | January 2023-March 2024
  Is sperm concentration different between men with HPV+ and HPV- semen samples?
Sperm motility in % of motile sperm | January 2023-March 2024
  Is sperm motility different between men with HPV+ and HPV- semen samples?
Fertilization rate | January 2023-March 2024
  Is the fertilization rate (number of fertilized oocytes) after IVF/ICSI treatment different between men with HPV+ and HPV- semen samples?
High quality embryos | January 2023-March 2024
  Is the number of high-quality embryos(number of blastocysts developed after fertilization) after IVF/ICSI treatment different between men with HPV+ and HPV- semen samples?

CONTACTS AND LOCATIONS:
Overall Officials: Randa Akouri, Ph.D., Principal Investigator — Sahlgrenska Academy, Gothenburg University, Gothenburg, Sweden
Locations (1):
- Department of Obstetrics and Gynecology, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Francis J, Karrberg C, Hermansson J, Lindh M, Ganidou S, Thurin-Kjellberg A, Lundin K, Akouri R, Tsiartas P. Seminal HPV detection: a pilot study comparing the preservation effectiveness and cost between a methanol-based solution and cryopreservation with liquid nitrogen. Asian J Androl. 2022 Sep-Oct;24(5):560-561. doi: 10.4103/aja202213. No abstract available. PMID 35488669
- [Derived] Francis J, Tsiartas P, Hreinsson J, Andersson M, Hermansson J, Gogas P, Papadimitriou T, Karrberg C, Brannstrom M, Akouri R. Semen HPV and IVF: insights from infection prevalence to embryologic outcomes. J Assist Reprod Genet. 2025 Jun;42(6):2053-2066. doi: 10.1007/s10815-025-03513-6. Epub 2025 May 22. PMID 40402400